CLINICAL TRIAL: NCT04699591
Title: Compassionate Use of Domperidone for Refractory Gastroparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jose Cocjin, MD, Physician, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12060310
Record Dates: First submitted 2020-12-28; First posted 2021-01-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: GERD; Gastroesophageal Reflux; Gastroparesis
Keywords: reflux; acid reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Study (Other): Receive domperidone 4 times a day, weight-dependent dose
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — Domperidone taken 4 times a day, dose based on body weight
  Other Names: Motilium; Motillium; Motinorm Costi; Nomit; Brulium; Molax

SUMMARY:
The purpose of this program is to allow the use of domperidone in children from 12 to 21 years of age with symptoms related to motility disorders and Gastroesophageal reflux disease (GERD) who have failed all the standard treatments for their condition.

DETAILED DESCRIPTION:
The following will need to be completed before the investigational treatment can begin:

* Your medical history will be reviewed to make sure domperidone is a safe option for treatment
* You will have a physical examination, including heart and breathing rates, blood pressure, height, weight, and an ECG. An ECG measures the electrical activity of the heart over a period of time. This is a non-invasive procedure and involves attaching sticky pads to your chest and recording your body's electrical activity on a machine. The study doctor/nurse will explain this in more detail to you.
* You will have up to 3 teaspoons of blood drawn through a needle in the arm to make sure it is safe for you to receive domperidone.
* You will have a pregnancy test if you are female.

If your tests results are acceptable, the following will happen to you:

* You will take domperidone 4 times per day. The dose will be calculated by your doctor according to your weight.
* Every two months for the first year, you will have a physical examination, including heart and breathing rates, blood pressure, height, weight, up to 3 teaspoons of blood drawn through a needle in your arm to measure blood levels, and an ECG.
* You will also have an ECG anytime there is an increase in the amount of domperidone you are taking.
* After the first year, if you are benefitting from taking domperidone you will have a physical examination, blood draw and ECG every six months until you stop taking domperidone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 12 - 21
3. Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.
4. Patients must have a comprehensive evaluation to eliminate other causes of their symptoms.
5. Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

   * increased prolactin levels
   * extrapyramidal side effects
   * breast changes
   * Cardiac arrhythmias including QT prolongation
   * There is a potential for increased risk of adverse events with the drugs and herbal supplements listed in the addendum (See Addendum on pages 24 and 25)
   * The coordinator/investigator will have a discussion with the family about the use of any of the medications and herbal supplements listed in the addendum to make sure they understand the increased risk of their use and the need to contact the investigators prior to using any of the listed medications and herbal supplements.

Exclusion Criteria:

1. History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.
2. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged Tc (QTc> 450 milliseconds for males, QTc>470 milliseconds for females).
3. Clinically significant electrolyte disorders.
4. Gastrointestinal hemorrhage or obstruction
5. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
6. Pregnant or breast feeding female
7. Known allergy to domperidone

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Change in disease severity | Up to 1 year
  refractory gastroparesis or GERD(Gastroesophageal Reflux Disease)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cocjin, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States